CLINICAL TRIAL: NCT03425461
Title: Phase I Study Combining an Anti-SEMA4D Antibody VX15/2503 With Checkpoint Inhibitors for Patients With Advanced Melanoma Who Have Progressed on Prior Anti-PD1/L1 Based Therapies
Brief Title: Anti-SEMA4D Monoclonal Antibody VX15/2503 With Nivolumab or Ipilimumab in Treating Patients With Stage III or IV Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Vaccinex Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-001570; NCI-2017-02395 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-001570 (Other: UCLA / Jonsson Comprehensive Cancer Center); P30CA016042 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-02-07 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (anti-SEMA4D VX15/2503, nivolumab) (Experimental): ARM A: Patients receive anti-SEMA4D monoclonal antibody VX15/2503 IV over 60 minutes and nivolumab IV over 30 minutes every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-SEMA4D Monoclonal Antibody VX15/2503; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacological Study
- Arm B (anti-SEMA4D VX15/2503, ipilimumab) (Experimental): Patients receive anti-SEMA4D monoclonal antibody VX15/2503 IV over 60 minutes and ipilimumab IV over 30 minutes every 21 days for courses 1-4, then receive anti-SEMA4D monoclonal antibody VX15/2503 every 28 days for subsequent courses for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-SEMA4D Monoclonal Antibody VX15/2503; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Anti-SEMA4D Monoclonal Antibody VX15/2503 — Given IV
  Other Names: moAb VX15/2503; VX15/2503
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm B (anti-SEMA4D VX15/2503, ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Arm A (anti-SEMA4D VX15/2503, nivolumab)
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized pilot phase I trial studies the side effects and best dose of anti-SEMA4D monoclonal antibody VX15/2503 when given together with nivolumab or ipilimumab in treating patients with stage III or IV melanoma. Monoclonal antibodies, such as anti-SEMA4D monoclonal antibody VX15/2503, nivolumab, and ipilimumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of the combination of anti-SEMA4D monoclonal antibody VX15/2503 (anti-SEMA4D VX15/2503) with nivolumab, or ipilimumab, in melanoma patients who have progressed on anti-PD1/L1 based checkpoint inhibitors.

II. To determine the recommended phase II dose and schedule of the combination of anti-SEMA4D VX15/2503 with nivolumab, or ipilimumab, in melanoma patients who have progressed on anti-PD1/L1 based checkpoint inhibitors.

SECONDARY OBJECTIVES:

I. Define the adverse event profile for the agent combinations and determine attribution (i.e. drug related adverse events [AEs]); II. To evaluate clinical response of patients treated with maximum tolerated dose (MTD) or maximum administered dose (MAD) of the combination of anti-SEMA4D with nivolumab, or ipilimumab.

III. To evaluate whether adding anti-SEMA4D to PD1 or CTLA-4 blockade can increase T-cell infiltration into tumors and whether change in T-cell infiltration is associated with response.

OUTLINE: This is a dose-escalation study of anti-SEMA4D monoclonal antibody VX15/2503. Patients are randomized to 1 of 2 arms.

ARM A: Patients receive anti-SEMA4D monoclonal antibody VX15/2503 intravenously (IV) over 60 minutes and nivolumab IV over 30 minutes every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive anti-SEMA4D monoclonal antibody VX15/2503 IV over 60 minutes and ipilimumab IV over 30 minutes every 21 days for courses 1-4, then receive anti-SEMA4D monoclonal antibody VX15/2503 every 28 days for subsequent courses for up to 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 2 years, every 6 months for 3 years, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed unresectable stage III or stage IV metastatic melanoma, who have not been previously treated with a SEMA4D antibody and have had prior anti-PD1/PDL1 inhibitors with documented progression; patient may have or not have prior anti-CTLA4 treatments
* Measurable disease per RECIST v. 1.1 criteria using imaging scans, or peripheral lesions that can be adequately documented with a picture and a ruler even if they do not meet RECIST criteria.
* Patients must have non-target lesion accessible for sequential biopsy (core needle biopsy or excision preferred, fine needle aspiration not eligible)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Women of child-bearing potential must have a negative serum pregnancy test within 24 hour of initiation of dosing and must agree to use an effective form of contraception during the study from the time of the negative pregnancy test up to 6 months after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive in conjunction with a barrier method, or a double barrier method. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for >= 1 year. Fertile men must also agree to use an effective method of birth control while on study drug and up to 6 months after the last dose of study drug
* Patients must have fully recovered from the effects of any major surgery or significant traumatic injury within 14 days of course 1 day 1 (C1D1)
* Absolute neutrophil count >= 1 X 10^9/L
* Hemoglobin (Hgb) > 8 g/dL
* Platelet count >= 75 X 10^9/L
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 X upper limit of normal (ULN) or < 5 X ULN in the presence of liver metastases
* Bilirubin =< 3 X ULN or < 5 X ULN in the presence of liver metastases
* Creatinine =< 3 X ULN or calculated creatinine clearance (CrCl) > 30 mL/min using Cockcroft- Gault formula
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements

Exclusion Criteria:

* Active secondary malignancy, unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the Medical Monitor.
* Investigational drug use within 28 days of C1D1
* Chemotherapy, targeted therapy, growth factors or radiation therapy within 14 days of C1D1
* Systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to registration
* History of any of the following toxicities associated with a prior immunotherapy:

  * Grade >= 3 immune mediated adverse event that was considered related to previous immunotherapy and required immune suppressive therapy. It is acceptable to allow patients with Grade 3 ophthalmologic immune-mediated events that improved to Grade 1 within 2 weeks after topical therapy only, and patients with Grade 3 endocrine immune-mediated events that did not experience symptoms lasting > 6 weeks and are not requiring > 7.5mg prednisone or equivalent per day.
  * Immune mediated adverse event that was considered related to previous immunotherapy and is still > grade 1 with immune suppressive therapy
  * • Any active immune-mediated adverse events requiring ongoing immune suppressive therapy (hormone replacement therapy is permitted).
* Patients with known active central nervous system (CNS) lesions are excluded (i.e., those with radiographically unstable, symptomatic lesions). However, patients treated with stereotactic therapy or surgery are eligible if they remain without evidence of disease progression in the brain for 14 days.
* Major surgery within 14 days of registration
* Has received a live vaccine within 28 days prior to registration
* A known active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness (human immunodeficiency virus [HIV] testing is not required), including patients who have an active infection requiring systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of anti-SEMA4D monoclonal antibody VX15/2503 determined by dose limiting toxicity assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 21 days
  Simple descriptive statistics will be used to summarize toxicities observed at each monitoring visit through the treatment and follow up period such as absolute neutrophil count), severity (by Toxicity Table) and nadir or maximum values for the laboratory measures, time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course. Baseline information (e.g. the extent of prior therapy) and demographic information will be presented, as well, to describe the patients treated in this pilot study.

SECONDARY OUTCOMES:
Antitumor activity assessed using tumor response | Up to 5 years
  Potential objective responses classifications (complete response [CR], partial response [PR] and stable disease) to this combinatorial immunotherapy will be defined and recorded following Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, immune related response criterion (irRC) and immune related RECIST (irRECIST) criteria.
Duration of response | From the time measurement criteria is met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented up to 5 years
Frequency of tumor measurements | Up to 5 years
Incidence of adverse events based on the Common Toxicity Criteria version 4.0 | Up to 2 years
  Adverse events will be tabulated by type, severity, and the frequency and proportion of subjects experiencing the event.
Response for in-transit metastasis | Up to 5 years
  Response will be assessed, taking the measurement from pictures with a built-in ruler.

OTHER OUTCOMES:
T cell Infiltration | Baseline and 4 weeks after treatment starts
  Will be analyzed using quantitative digital pathology.
T cell receptor (TCR) clonality in tumors | Baseline and 4 weeks after treatment starts
  Will analyze TCR clonality by deep sequencing the TCR Vbeta complementarity-determining region (CDR) region using the ImmunoSeq assay from Adaptive Biotech.
Tumor immune microenvironment | Baseline and 4 weeks after treatment starts
  Will be assessed using immunohistochemistry and analyzed using quantitative digital pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No